CLINICAL TRIAL: NCT00867685
Title: A Phase I, Randomized, Open Label, 2-Way Crossover Study in Healthy Subjects to Assess the Relative Bioavailability of AZD2624 (Tablet Versus Liquid Suspension) Followed by an Additional Period to Assess the Food Effect on the Tablet
Brief Title: Phase I 2-Way Crossover Study to Assess Relative BA of Tablet Versus Liquid Suspension and Food Effect on Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Smith, MD, PhD, Senior Medical ScienceDirector Emerging Neuroscience, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D0970C00008
Record Dates: First submitted 2009-03-18; First posted 2009-03-24 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — 3-((methylsulfonyl)amino)-2-phenyl-N-(1-phenylpropyl)quinolin-4-carboxamide

ARMS (3):
- Treatment A (Experimental): Single oral dose of 40 mg AZD2624 liquid suspension in a fasted state.
  Interventions: Drug: AZD2624
- Treatment B (Experimental): Single oral dose of 40 mg (2x20mg tablets)AZD2624 in a fasted state.
  Interventions: Drug: AZD2624
- Treatment C (Experimental): Single oral dose of 40 mg (2x20mg tablets) in a fed state.
  Interventions: Drug: AZD2624

INTERVENTIONS:
Drug: AZD2624 — Single dose of 40 mg AZD2624 liquid suspension, PO
  Arms: Treatment A
Drug: AZD2624 — Single dose of 40 mg AZD 2624 (2x20mg tablets), PO
  Arms: Treatment B; Treatment C

SUMMARY:
The purpose of this study is to compare the liquid suspension form of AZD 2624 to a tablet form of the same drug. This study will also study the effect of food on the tablet form of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers

Exclusion Criteria:

* Donation of plasma or blood products within one month of of screening
* Clinically relevant abnormalities in physical examination, vital signs,ECG, clinical chemistry, hematology, or urinalysis.
* Previous participation in an AD2624 study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Serial blood draws will be used to measure the plasma levels of AZD2624 for the liquid suspension and the tablet formulation in a fed and fasted state. | Seventeen blood draws will be collected during each treatment period for a total of 51 samples for the study.

SECONDARY OUTCOMES:
Safety will be measured by the collection of AEs, ECGs, physical exams, and vital signs. | Subjects inquiry on AE daily, ECGs collected at 2 timepoints each period, clinical labs collected at 3 timepoints each period, physical exams completed 3 timepoints each period, and vital signs collected each day of each period

CONTACTS AND LOCATIONS:
Overall Officials: Sylvan Hurewitz, MD, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, US
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States